CLINICAL TRIAL: NCT04856696
Title: Clinical Application of Non-invasive Preimplantation Genetic Testing for Aneuploidies
Brief Title: Clinical Application of Non-invasive PGT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Sofiva Genomics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Principal Investigator, Assistant professor, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KSVGH20-CT12-16
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Genetic Testing
Keywords: PGT; PGT-A; non-invasive PGT-A; embryo biopsy; spent media; cell free DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined non-invasive PGT-A & PGT-A (Experimental): Infertility women who underwent both non-invasive PGT-A and PGT-A
  Interventions: Diagnostic Test: PGT-A; Diagnostic Test: non-invasive PGT-A
- non-invasive PGT-A (Experimental): Infertility women who underwent non-invasive PGT-A only
  Interventions: Diagnostic Test: non-invasive PGT-A
- PGT-A (Active Comparator): Infertility women who underwent PGT-A only
  Interventions: Diagnostic Test: PGT-A

INTERVENTIONS:
Diagnostic Test: PGT-A — trophectoderm biopsy in blastocyst stage for euploidy testing using next generation sequencing platform
  Arms: PGT-A; combined non-invasive PGT-A & PGT-A
Diagnostic Test: non-invasive PGT-A — cell-free DNA collected from spent culture media for euploidy testing using next generation sequencing platform
  Arms: combined non-invasive PGT-A & PGT-A; non-invasive PGT-A

SUMMARY:
The study aims to investigate the difference of in vitro fertilization (IVF) outcomes among non-invasive PGT-A, PGT-A and combined non-invasive PGT-A and PGT-A.

DETAILED DESCRIPTION:
Background Chromosome abnormality is a leading cause of implantation failure and miscarriage. Chromosome abnormality increases with age, resulting in reduced pregnancy rate. Nowadays, preimplantation genetic testing for aneuploidies (PGT-A) could be used for detection of aneuploidy. However, PGT-A needs embryo biopsy which is invasive and may cause embryo damage. It was found that cell free DNA could be isolated from culture media. The cell free DNA from culture media also could be used to detect embryo ploidy, called non-invasive PGT-A.

Objective The study aims to investigate the difference of in vitro fertilization (IVF) outcomes among non-invasive PGT-A, PGT-A and combined non-invasive PGT-A and PGT-A. Another aim of this study is to check the concordance rate between non-invasive PGT-A and PGT-A.

Methods The prospective cohort study will be performed at the reproductive medical center of Kaohsiung Veterans General Hospital, in Kaohsiung, Taiwan. Participants who plan to receive an IVF cycle and preimplantation genetic testing for aneuploidies will be enrolled in this study. The investigators will divide the participants into 3 groups: (1) combined non-invasive PGT-A and PGT-A; (2) PGT-A; (3) non-invasive PGT-A. Basal characteristics, infertility history, ovarian reserve and embryo development of the three groups will be recorded. The samples will be detected ploidy by using next generation sequencing (NGS). Then, the investigators will choose embryo to transfer according to the embryo ploidy and follow the pregnancy outcomes after embryo transfer.

Outcome

1. Concordance rate between non-invasive PGT-A and PGT-A
2. The relationship between morphological grade and ploidy of non-invasive PGT-A
3. IVF outcomes among non-invasive PGT-A, PGT-A and combined non-invasive PGT-A and PGT-A

ELIGIBILITY:
Inclusion Criteria:

* Infertile women who undergo IVF with PGT
* BMI:18~30 kg/m2

Exclusion Criteria:

* Primary ovarian insufficiency
* Congenital uterine anomaly
* Severe male infertility (azoospermia)
* One of the couples with chromosome abnormality
* Malignancy

Ages: 30 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | through study completion, an average of 1.5 year
  continuous presence of a fetal heartbeat over 12 weeks of a pregnancy

SECONDARY OUTCOMES:
Clinical pregnancy rate | through study completion, an average of 1.5 year
  the presence of a fetal heartbeat at 6-7 weeks of a pregnancy
Miscarriage rate | through study completion, an average of 1.5 year
  pregnancy loss before 24 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fesahat F, Montazeri F, Hoseini SM. Preimplantation genetic testing in assisted reproduction technology. J Gynecol Obstet Hum Reprod. 2020 May;49(5):101723. doi: 10.1016/j.jogoh.2020.101723. Epub 2020 Feb 26. PMID 32113002
- [Background] Sciorio R, Dattilo M. PGT-A preimplantation genetic testing for aneuploidies and embryo selection in routine ART cycles: Time to step back? Clin Genet. 2020 Aug;98(2):107-115. doi: 10.1111/cge.13732. Epub 2020 Apr 6. PMID 32141057
- [Background] Homer HA. Preimplantation genetic testing for aneuploidy (PGT-A): The biology, the technology and the clinical outcomes. Aust N Z J Obstet Gynaecol. 2019 Apr;59(2):317-324. doi: 10.1111/ajo.12960. Epub 2019 Feb 27. PMID 30811595
- [Background] Fragouli E, Munne S, Wells D. The cytogenetic constitution of human blastocysts: insights from comprehensive chromosome screening strategies. Hum Reprod Update. 2019 Jan 1;25(1):15-33. doi: 10.1093/humupd/dmy036. PMID 30395265
- [Background] Sullivan-Pyke C, Dokras A. Preimplantation Genetic Screening and Preimplantation Genetic Diagnosis. Obstet Gynecol Clin North Am. 2018 Mar;45(1):113-125. doi: 10.1016/j.ogc.2017.10.009. PMID 29428279
- [Background] Rubio C, Navarro-Sanchez L, Garcia-Pascual CM, Ocali O, Cimadomo D, Venier W, Barroso G, Kopcow L, Bahceci M, Kulmann MIR, Lopez L, De la Fuente E, Navarro R, Valbuena D, Sakkas D, Rienzi L, Simon C. Multicenter prospective study of concordance between embryonic cell-free DNA and trophectoderm biopsies from 1301 human blastocysts. Am J Obstet Gynecol. 2020 Nov;223(5):751.e1-751.e13. doi: 10.1016/j.ajog.2020.04.035. Epub 2020 May 26. PMID 32470458
- [Background] Rubio C, Rienzi L, Navarro-Sanchez L, Cimadomo D, Garcia-Pascual CM, Albricci L, Soscia D, Valbuena D, Capalbo A, Ubaldi F, Simon C. Embryonic cell-free DNA versus trophectoderm biopsy for aneuploidy testing: concordance rate and clinical implications. Fertil Steril. 2019 Sep;112(3):510-519. doi: 10.1016/j.fertnstert.2019.04.038. Epub 2019 Jun 11. PMID 31200971
- [Background] Leaver M, Wells D. Non-invasive preimplantation genetic testing (niPGT): the next revolution in reproductive genetics? Hum Reprod Update. 2020 Jan 1;26(1):16-42. doi: 10.1093/humupd/dmz033. PMID 31774124
- [Background] Kuznyetsov V, Madjunkova S, Abramov R, Antes R, Ibarrientos Z, Motamedi G, Zaman A, Kuznyetsova I, Librach CL. Minimally Invasive Cell-Free Human Embryo Aneuploidy Testing (miPGT-A) Utilizing Combined Spent Embryo Culture Medium and Blastocoel Fluid -Towards Development of a Clinical Assay. Sci Rep. 2020 Apr 29;10(1):7244. doi: 10.1038/s41598-020-64335-3. PMID 32350403
- [Background] Liang B, Gao Y, Xu J, Song Y, Xuan L, Shi T, Wang N, Hou Z, Zhao YL, Huang WE, Chen ZJ. Raman profiling of embryo culture medium to identify aneuploid and euploid embryos. Fertil Steril. 2019 Apr;111(4):753-762.e1. doi: 10.1016/j.fertnstert.2018.11.036. Epub 2019 Jan 22. PMID 30683589
- [Background] Jiao J, Shi B, Sagnelli M, Yang D, Yao Y, Li W, Shao L, Lu S, Li D, Wang X. Minimally invasive preimplantation genetic testing using blastocyst culture medium. Hum Reprod. 2019 Jul 8;34(7):1369-1379. doi: 10.1093/humrep/dez075. PMID 31251795
- [Background] Huang L, Bogale B, Tang Y, Lu S, Xie XS, Racowsky C. Noninvasive preimplantation genetic testing for aneuploidy in spent medium may be more reliable than trophectoderm biopsy. Proc Natl Acad Sci U S A. 2019 Jul 9;116(28):14105-14112. doi: 10.1073/pnas.1907472116. Epub 2019 Jun 24. PMID 31235575
- [Background] Fang R, Yang W, Zhao X, Xiong F, Guo C, Xiao J, Chen L, Song X, Wang H, Chen J, Xiao X, Yao B, Cai LY. Chromosome screening using culture medium of embryos fertilised in vitro: a pilot clinical study. J Transl Med. 2019 Mar 8;17(1):73. doi: 10.1186/s12967-019-1827-1. PMID 30849973
- [Background] Vera-Rodriguez M, Diez-Juan A, Jimenez-Almazan J, Martinez S, Navarro R, Peinado V, Mercader A, Meseguer M, Blesa D, Moreno I, Valbuena D, Rubio C, Simon C. Origin and composition of cell-free DNA in spent medium from human embryo culture during preimplantation development. Hum Reprod. 2018 Apr 1;33(4):745-756. doi: 10.1093/humrep/dey028. PMID 29471395
- [Background] Belandres D, Shamonki M, Arrach N. Current status of spent embryo media research for preimplantation genetic testing. J Assist Reprod Genet. 2019 May;36(5):819-826. doi: 10.1007/s10815-019-01437-6. Epub 2019 Mar 21. PMID 30895497
- [Background] Farra C, Choucair F, Awwad J. Non-invasive pre-implantation genetic testing of human embryos: an emerging concept. Hum Reprod. 2018 Dec 1;33(12):2162-2167. doi: 10.1093/humrep/dey314. PMID 30357338
- [Background] Xu J, Fang R, Chen L, Chen D, Xiao JP, Yang W, Wang H, Song X, Ma T, Bo S, Shi C, Ren J, Huang L, Cai LY, Yao B, Xie XS, Lu S. Noninvasive chromosome screening of human embryos by genome sequencing of embryo culture medium for in vitro fertilization. Proc Natl Acad Sci U S A. 2016 Oct 18;113(42):11907-11912. doi: 10.1073/pnas.1613294113. Epub 2016 Sep 29. PMID 27688762
- [Background] Shamonki MI, Jin H, Haimowitz Z, Liu L. Proof of concept: preimplantation genetic screening without embryo biopsy through analysis of cell-free DNA in spent embryo culture media. Fertil Steril. 2016 Nov;106(6):1312-1318. doi: 10.1016/j.fertnstert.2016.07.1112. Epub 2016 Aug 24. PMID 27565258
- [Background] Youssef MM, Mantikou E, van Wely M, Van der Veen F, Al-Inany HG, Repping S, Mastenbroek S. Culture media for human pre-implantation embryos in assisted reproductive technology cycles. Cochrane Database Syst Rev. 2015 Nov 20;2015(11):CD007876. doi: 10.1002/14651858.CD007876.pub2. PMID 26585317